CLINICAL TRIAL: NCT05189418
Title: Sleep-time Blood Pressure Determined by Home and Ambulatory Monitoring as Potential Prognostic Factor for Chronic Kidney Disease (CKD) Progression, Mortality, and Cardiovascular Morbidity in Patients With Advanced CKD
Brief Title: Sleep-time Blood Pressure and Risk of CKD Progression
Acronym: SLEEP-BP-CKD
Status: Completed | Type: Observational
Sponsor: University of Vigo (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Servicio Gallego de Salud (Other Government); University of Texas at Austin (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ramon C. Hermida, Full Professor, Director of Bioengineering & Chronobiology Labs, University of Vigo
Other Study IDs: SLEEP-BP-CKD; 2021-002585-41 (EudraCT Number); 2021/451 (Registry Identifier: Committee of Ethics in Investigation of Galicia)
Record Dates: First submitted 2021-12-23; First posted 2022-01-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: Ambulatory blood pressure monitoring; Home blood pressure monitoring; Chronic kidney disease; Cardiovascular risk; Sleep-time blood pressure; Blood pressure dipping
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring (ABPM) — Periodic (quarterly) 48h ABPM evaluation during follow-up
Device: Home blood pressure monitoring (HBPM) — Periodic (monthly) 7-day HBPM, both during awake and sleep spans, during follow-up

SUMMARY:
The SLEEP-BP-CKD Study has been designed to specifically test the following primary hypotheses:

(i) Specific ABPM-derived parameters, in particular the asleep SBP mean and/or the sleep-time relative SBP decline, are significant prognostic markers of deterioration of kidney function and progression towards ESKD, as well as of the risk of all-cause mortality and major CVD events, in high-risk patients with stage G3b-G4 CKD.

(ii) Changes during follow-up in specific ABPM-derived parameters, in particular the increase of the asleep SBP mean and/or decrease of the sleep-time relative SBP decline towards the non-dipper/riser 24h SBP pattern, are significant prognostic markers of deterioration of kidney function and progression towards ESKD, as well as of the risk of all-cause mortality and major CVD events, in high-risk patients with stage G3b-G4 CKD.

A novelty of the SLEEP-BP-CKD Study is the incorporation of clinical-grade wearable digital technology to monitor both wake-time and sleep-time BP at home in a subgroup (up to 200) of the total sample; this procedure will provide added useful information to test the following additional hypotheses:

(iii) The HBPM self-assessment procedure to obtain BP measurements both during wake-time and sleep-time spans provides reliable data to be used either individually or jointly with periodic ABPM as added potential prognostic marker of deterioration of kidney function and progression towards ESKD, as well as of the risk of all-cause mortality and major CVD events, in high-risk patients with stage G3b-G4 CKD.

(iv) The sleep-time BP measurements obtained by HBPM self-assessment and their changes during follow-up are better correlated, compared with wake-time OBPM or wake-time HBPM, to eGFR and albuminuria (measured by the albumin/creatinine ratio) and their changes during follow-up, respectively.

(v) The HBPM self-assessment procedure to obtain BP measurements both during wake-time and sleep-time spans increases patient adherence/compliance to prescribed treatment from baseline.

The scheduled periodic patient BP assessments during follow-up with OBPM, HBPM, 48h ABPM, along with laboratory urine and blood test data will further allow evaluating and comparing the changes from baseline in all these clinically relevant variables as potential markers for risk of progression towards ESKD, all-cause mortality, and/or CVD morbidity.

DETAILED DESCRIPTION:
Hypertension is very common in patients with chronic kidney disease (CKD); its prevalence increases with diminished estimated glomerular filtration rate (eGFR), reaching an estimated 86% in patients with end-stage kidney disease (ESKD). On the other hand, hypertension leads to kidney and other target-organ damage, through its burden of mechanical and oxidative stress on vascular walls.

As in the past, current hypertension guidelines continue to recommend wake-time office blood pressure (BP) measurement (OBPM) as the primary mode of diagnosing hypertension and establishing therapeutic goals. Nonetheless, many of them now advocate ambulatory BP (ABP) monitoring (ABPM) of adult patients to confirm the OBPM-based diagnosis of hypertension because of the well-documented significantly better value of ABPM-derived parameters relative to wake-time OBPM in prognosticating cardiovascular disease (CVD) risk, a relevant finding also well documented in patients with CKD. Unfortunately, ABPM is seldom applied in clinical practice, and when it is, there is no consensus as of yet exactly how to properly apply it, e.g., how frequent to sample BP and for how long, and also what parameter(s) to use for making accurate diagnosis. Most guidelines propose around-the-clock ABPM to derive for diagnostic purpose either the 24h or the "daytime" systolic (SBP) and diastolic BP (DBP) means that typically are defined according to fixed clock time durations established by default by the manufacturers of the measuring devices or set a priori by investigators as opposed to biologically meaningful ones based on the actual clock times of the beginning and end of the activity and sleep spans of each patient to derive accurate individualized awake and asleep BP means and dipping pattern.

Contrary to the recommendation of the most recently published hypertension guidelines to rely on the "daytime" or 24h ABP means to diagnose hypertension when ABPM is performed, multiple prospective outcome trials and meta-analyses substantiate CVD events are much better predicted by the asleep BP mean. CVD risk is additionally predicted by an attenuated sleep-time relative SBP decline - non-dipper (sleep-time relative SBP decline <10%) or riser (sleep-time relative SBP decline <0%) 24h SBP profile. Thus, the elevated asleep SBP mean and blunted sleep-time relative SBP decline (non-dipping) constitute joint significant CVD risk factors, independent of the wake-time OBPM or the awake or 24h ABP means. The importance of the asleep SBP mean for making the diagnosis and prognosis of CVD risk is exemplified by a meta-analysis of the original databases of nine cohorts representing in total 13,844 hypertensive patients. It found that the wake-time office SBP as well as ABPM-derived awake and asleep SBP means were all significantly associated with elevated CVD risk when each variable was analyzed individually; however, when all three SBP measurements were simultaneously included into the survival model, only the asleep SBP mean remained as the independent BP-derived predictor of CVD events.

The differential relevance of several ABPM-derived parameters, compared with the wake-time OBPM, as potential risk markers of CVD morbidity and mortality has been further assessed in the thus far largest reported primary care-based ABPM-based investigation, the Hygia Project, established in 2007 as a multicenter research network - currently comprised of 40 primary care facilities and 292 clinical investigators - designed to incorporate ABPM as routine procedure to diagnose and manage hypertension, assess efficacy of BP-lowering treatment, and evaluate patient CVD and other medical risks. Between 2008 and 2018, participating primary-care physicians - properly trained and certified in the proper application of ABPM and the conduct of procedures of the investigative protocol - referred in total 21,963 primary care patients for 48h ABPM annually, or more frequently when the ABP of treated hypertensive patients remained uncontrolled, i.e., ≥135/85 or ≥120/70 mmHg for, respectively, the awake and asleep SBP/DBP means and those having compelling clinical conditions of elevated CVD risk, including diabetes, CKD, and past major CVD event. During the median follow-up of 6.3 years, 1,830 individuals experienced the main CVD-outcome of CVD death, myocardial infarction, coronary revascularization, heart failure, ischemic stroke, or hemorrhagic stroke. Corroborating and extending previously reported findings - based upon an initial analysis of the data of the Hygia Project cohort of 18,078 individuals that had been recruited up to 2015 - Cox proportional-hazard analyses revealed the asleep SBP mean to be the most significant single BP marker of CVD risk, independent of absence/presence of hypertension therapy at baseline, upon-waking vs. at-bedtime treatment-time, diagnosis of influential morbidities of diabetes or CKD, age, and sex. The joint contribution with the asleep SBP mean to CVD risk was significant only for diminished sleep-time relative SBP decline but not for the wake-time OBPM or the awake or 24h ABP means, such that at any given asleep SBP level, non-dipper individuals showed significantly greater CVD risk than did dipper ones.

A blunted sleep-time BP decline, which is characteristic of the non-dipper/riser 24h BP pattern, is common in patients with CKD. Nonetheless, the reported prevalence of sleep-time hypertension and non-dipping in CKD in different studies is highly inconsistent and, thus, its exact prevalence and associated potential clinical relevance are uncertain. Among other factors, this might be due to differences in the studied populations (treated or untreated patients at differing stages of CKD), relatively small sample sizes, definition of awake and asleep periods by arbitrary fixed clock-hour spans, and frequent reliance only on a single, low-reproducible, 24h ABPM evaluation per participant. Moreover, most previous investigations have evaluated the 24h BP pattern of patients with CKD exclusive of proper comparison to those without CKD.

Several prospective studies have investigated the prognostic value of the features of the 24h BP pattern determined by around-the-clock ABPM for prediction of the development and progression of CKD. Some of these studies, in particular, have found sleep-time hypertension and the non-dipper/rising BP pattern to be predictors of the development and progression of albuminuria, worsening proteinuria, decline in eGFR, and progression to ESKD.

The MAPEC Study investigated the prognostic value of OBPM and ABP to predict new-onset CKD and whether risk reduction might be associated with progressive treatment-induced decrease of wake-time OBPM or ABPM-determined awake or asleep BP means. The authors prospectively evaluated 2,763 individuals without CKD and with baseline ABP ranging from normotension to hypertension. Upon recruitment and annually (or more frequently if hypertension treatment was adjusted based on ABP targets) thereafter, BP and physical activity (wrist actigraphy) were simultaneously monitored for 48h to accurately derive individualized awake and asleep BP means. During a 5.9-year median follow-up, 404 participants developed CKD. CKD risk was greater with progressively higher asleep SBP mean and lower sleep-time relative SBP decline, i.e., more non-dipper BP pattern. The asleep SBP mean was indeed the most significant predictor of CKD in a Cox proportional-hazard model adjusted for age, diabetes, serum creatinine, urinary albumin, previous CVD event, and hypertension treatment-time, i.e., upon-awakening vs. at-bedtime (per 1-SD elevation, hazard ratio 1.44, [95%CI: 1.31-1.56], P<0.001). Wake-time OBPM and awake or 48h ABP means lost their predictive value when corrected by the asleep SBP mean. Analyses of BP changes during follow-up revealed 27% reduction in the risk of CKD per 1-SD decrease in asleep SBP mean, independent of changes in wake-time OBPM or awake ABP mean. In conclusion, sleep-time SBP is a highly significant independent prognostic marker for CKD. Alteration of sleep-time SBP regulation, i.e., increase in asleep SBP mean or blunted sleep-time relative SBP decline, seems to precede, rather than follow, the development of CKD. Furthermore, the progressive treatment-induced decrease of asleep SBP mean, a potential therapeutic target requiring around-the-clock ABPM patient evaluation, might be a significant method for establishing an effective therapeutic regimen to reduce or avert the risk for CKD. Despite these collective findings from ABPM-based clinical trials, current models for predicting the development and progression of CKD either do not include BP as a relevant covariate or rely solely on the wake-time OBPM.

On the other hand, home BP monitoring (HBPM) has been advocated as the preferred method for out-of-office BP assessment by current guidelines to corroborate the diagnosis of hypertension based on wake-time OBPM. This preference seems to be based on some apparent advantages over ABPM, including HBPM being widely used, cost-efficient, and well accepted by hypertensive patients for long-term BP evaluation and potential improvement of compliance with hypertension treatment. The major shortcoming of conventional HBPM devices of the past is that BP measurement could not be programmed and, accordingly, they were not capable of measuring BP during sleep.

Recent advances in self-monitoring device technology have enabled measurement of BP during sleep. The currently available sleep-time HBPM devices provide automatic triggering of a few asleep BP measurements. In particular, the NightView (Omron Healthcare, HEM9601T-E3) is a light (110 g) wrist type HBPM device that, in addition to customary wake-time BP measurements (triggered upon demand by the patient), it also automatically takes BP measurements during sleep. The NightView device has been clinically validated for use in the sitting and in supine position (with palm placed sideways, upwards, and downwards) according to the ANSI/AAMI/ISO81060-2:2013 protocol and it passed all criteria.

The primary objectives of the study are:

1. To prospectively evaluate the prognostic value of sleep-time BP assessed by HBPM and ABPM, as well as its treatment-induced changes during follow-up, as potential makers for progression of CKD.
2. To prospectively evaluate the prognostic value of sleep-time BP assessed by HBPM and ABPM, as well as its treatment-induced changes during follow-up, as potential makers for total and CVD mortality in patients with advanced CKD.
3. To prospectively evaluate the prognostic value of sleep-time BP assessed by HBPM and ABPM, as well as its treatment-induced changes during follow-up, as potential makers for CVD morbidity in patients with advanced CKD.
4. To evaluate, for all of the primary objectives listed above, the potential influence of other HBPM and ABPM-determined parameters of interest as well as their treatment-induced changes during follow-up, including (but not limited to) the sleep-time relative SBP decline (measure of 24h SBP dipping), 48h and awake BP means, measurements of BP variability, ambulatory arterial stiffness index (AASI), morning BP surge, pre-awakening BP surge, and sleep-time BP fall.
5. After assessment of the prognostic value of all potential significant covariates, to develop a risk score system for individualized stratification of patients with advanced CKD.

Required sample size calculation:

If each patient would be evaluated by 48h ABPM only twice, i.e., at baseline and after follow-up, we will obtain two values of each potential prognostic BP variable, but only one of the change in those variables during follow-up. Under this hypothetical situation, at the two-sided a level of 5% and with a power of 80%, 450 participants providing all required information would make possible the detection of a difference of >30% in the incidence of the composite outcome variable after a median follow-up of >1.5 years in patients divided according to each tested prognostic factor or its change during follow-up (e.g., normal/controlled vs. elevated sleep-time SBP mean, dipper vs. non-dipper, etc.). However, by protocol design, each participant will be scheduled for multiple 48h ABPM assessment, i.e., at baseline and then every 3 months during follow up. For a median follow-up of 1.5 years from baseline, participants might provide up to 7 ABPM profiles, with the corresponding 6 values of changes in BP parameters from baseline to each of the quarterly 48h ABPM assessments. Accordingly, due to the unique design of this protocol, at the two-sided a level of 5% and with a power of 80%, a maximum of 160 participants would make possible the detection of a difference of >30% in the incidence of the composite outcome variable after a median follow-up of >1.5 years in patients divided according to each tested prognostic factor or its change during follow-up. Recruitment of an additional up to 20% of the target sample (thus 192 patients in total) will be sought to cover possible dropouts and/or lack of the required 1-year minimum follow-up per participant. These sample size requirements might need to be recalculated as a function of the actual incidence of events (for the defined composite renal+CVD primary outcome) documented during the first year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years.
2. Wrist circumference between 13.5 and 21.5 cm to enable proper use of the NightView HBPM device (only for those who might use it).
3. Upon recruitment have moderate to severely decreased eGFR, i.e., stages G3b (eGFR 30-44 ml/min/1.73 m2) or G4 (eGFR 15-29 ml/min/1.73 m2).
4. Agreement to adhere lifestyle considerations (routine of daytime activity and nighttime sleep) and mandates (e.g., wearing of NightView and ABPM devices) of the investigative protocol.
5. Provision of written informed consent to participate into the study.

Exclusion Criteria:

1. Pregnancy.
2. History of alcoholism or narcotic addiction within the last two years.
3. Night, rotating shift-work employment, or frequent transmeridian travel.
4. Previous history of a systemic autoimmune disease or AIDS.
5. Evidence of a secondary form of hypertension, including coarctation of the aorta, hyperaldosteronism, renal artery stenosis, or pheochromocytoma.
6. Severe cardiac disease (unstable angina pectoris, unstable heart failure, life-threatening arrhythmia, and atrial fibrillation). Previous CVD events will not be exclusionary if full physical and work activities are maintained.
7. Any surgical or medical condition which might alter the absorption, distribution, metabolism, or excretion of any medication, or, at the discretion of the investigator, might place the subject at higher medical risk from his/her participation in the study, or is likely to prevent the subject from complying with the requirements of the study or completing the trial period.
8. History of any malignancy within the past five years, including leukemia and lymphoma (but not basal cell skin cancer), or any other severe disease if involving life-threatening risk.
9. Inability to communicate and comply with all study requirements.
10. Intolerance to or unacceptance of ABPM or HBPM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who upon recruitment have moderate to severely decreased eGFR, i.e., stages G3b (eGFR 30-44 ml/min/1.73 m2) or G4 (eGFR 15-29 ml/min/1.73 m2).
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
CKD-progression | 2 years
  Composite of 30% decrease in eGFR, 30% increase in albuminuria, or ESKD
CVD-outcome | 2 years
  Composite of CVD death, myocardial infarction, coronary revascularization, heart failure, ischemic stroke, and hemorrhagic stroke.
Renal+CVD-outcome | 2 years
  Composite of 30% decrease in eGFR, 30% increase in albuminuria, ESKD, all-cause mortality, or major CVD event

SECONDARY OUTCOMES:
Coronary events | 2 years
  Composite of CVD death, myocardial infarction, and coronary revascularization.
Cardiac events | 2 years
  Composite of coronary events and heart failure.
Stroke | 2 years
  Composite of ischemic stroke and hemorrhagic stroke.
Total CVD events | 2 years
  Composite of CVD death, myocardial infarction, coronary revascularization, heart failure, ischemic stroke, hemorrhagic stroke, transient ischemic attack, angina pectoris, or peripheral artery disease.
Minor CVD events | 2 years
  Composite of angina pectoris, peripheral artery disease, thrombotic occlusion of the retinal artery, and transient ischemic attack.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Principal Investigator — University of Vigo; Michael H Smolensky, PhD, Principal Investigator — University of Texas at Austin; Sherine El-Toukhy, PhD, Principal Investigator — National Institute on Minority Health and Health Disparities (NIMHD); Keith C Norris, PhD, Principal Investigator — University of California, Los Angeles
Locations (10):
- Spain (10):
  - CS A Estrada, A Estrada, Pontevedra
  - Centro de Salud de A Doblada, Vigo, Pontevedra
  - Policlinico Vigo SA - POVISA, Vigo, Pontevedra
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro de Salud de Bembrive, Vigo, Pontevedra
  - Centro de Salud de Lavadores, Vigo, Pontevedra
  - Centro de Salud de Sardoma, Vigo, Pontevedra
  - CS Teis, Vigo, Pontevedra
  - Bioengineering & Chronobilogy Labs., University of Vigo, Vigo, Pontevedra
  - CS San Roque, Vilagarcía de Arousa, Pontevedra

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asayama K, Fujiwara T, Hoshide S, Ohkubo T, Kario K, Stergiou GS, Parati G, White WB, Weber MA, Imai Y; International Expert Group of Nocturnal Home Blood Pressure. Nocturnal blood pressure measured by home devices: evidence and perspective for clinical application. J Hypertens. 2019 May;37(5):905-916. doi: 10.1097/HJH.0000000000001987. PMID 30394982
- [Background] Cheng D, Tang Y, Li H, Li Y, Sang H. Nighttime blood pressure decline as a predictor of renal injury in patients with hypertension: a population-based cohort study. Aging (Albany NY). 2019 Jul 5;11(13):4310-4322. doi: 10.18632/aging.101873. PMID 31276448
- [Background] Coresh J, Turin TC, Matsushita K, Sang Y, Ballew SH, Appel LJ, Arima H, Chadban SJ, Cirillo M, Djurdjev O, Green JA, Heine GH, Inker LA, Irie F, Ishani A, Ix JH, Kovesdy CP, Marks A, Ohkubo T, Shalev V, Shankar A, Wen CP, de Jong PE, Iseki K, Stengel B, Gansevoort RT, Levey AS. Decline in estimated glomerular filtration rate and subsequent risk of end-stage renal disease and mortality. JAMA. 2014 Jun 25;311(24):2518-2531. doi: 10.1001/jama.2014.6634. PMID 24892770
- [Background] Coresh J, Heerspink HJL, Sang Y, Matsushita K, Arnlov J, Astor BC, Black C, Brunskill NJ, Carrero JJ, Feldman HI, Fox CS, Inker LA, Ishani A, Ito S, Jassal S, Konta T, Polkinghorne K, Romundstad S, Solbu MD, Stempniewicz N, Stengel B, Tonelli M, Umesawa M, Waikar SS, Wen CP, Wetzels JFM, Woodward M, Grams ME, Kovesdy CP, Levey AS, Gansevoort RT; Chronic Kidney Disease Prognosis Consortium and Chronic Kidney Disease Epidemiology Collaboration. Change in albuminuria and subsequent risk of end-stage kidney disease: an individual participant-level consortium meta-analysis of observational studies. Lancet Diabetes Endocrinol. 2019 Feb;7(2):115-127. doi: 10.1016/S2213-8587(18)30313-9. Epub 2019 Jan 8. PMID 30635225
- [Background] Gabbai FB, Rahman M, Hu B, Appel LJ, Charleston J, Contreras G, Faulkner ML, Hiremath L, Jamerson KA, Lea JP, Lipkowitz MS, Pogue VA, Rostand SG, Smogorzewski MJ, Wright JT, Greene T, Gassman J, Wang X, Phillips RA; African American Study of Kidney Disease and Hypertension (AASK) Study Group. Relationship between ambulatory BP and clinical outcomes in patients with hypertensive CKD. Clin J Am Soc Nephrol. 2012 Nov;7(11):1770-6. doi: 10.2215/CJN.11301111. Epub 2012 Aug 30. PMID 22935847
- [Background] International Society for Chronobiology; American Association of Medical Chronobiology and Chronotherapeutics; Spanish Society of Applied Chronobiology, Chronotherapy, and Vascular Risk; Spanish Society of Atherosclerosis; Romanian Society of Internal Medicine; Hermida RC, Smolensky MH, Ayala DE, Portaluppi F. 2013 ambulatory blood pressure monitoring recommendations for the diagnosis of adult hypertension, assessment of cardiovascular and other hypertension-associated risk, and attainment of therapeutic goals. Chronobiol Int. 2013 Apr;30(3):355-410. doi: 10.3109/07420528.2013.750490. PMID 23517220
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Sleep-Time Ambulatory BP Is an Independent Prognostic Marker of CKD. J Am Soc Nephrol. 2017 Sep;28(9):2802-2811. doi: 10.1681/ASN.2016111186. Epub 2017 Apr 28. PMID 28455314
- [Background] Hermida RC, Crespo JJ, Otero A, Dominguez-Sardina M, Moya A, Rios MT, Castineira MC, Callejas PA, Pousa L, Sineiro E, Salgado JL, Duran C, Sanchez JJ, Fernandez JR, Mojon A, Ayala DE; Hygia Project Investigators. Asleep blood pressure: significant prognostic marker of vascular risk and therapeutic target for prevention. Eur Heart J. 2018 Dec 14;39(47):4159-4171. doi: 10.1093/eurheartj/ehy475. PMID 30107515
- [Background] Ida T, Kusaba T, Kado H, Taniguchi T, Hatta T, Matoba S, Tamagaki K. Ambulatory blood pressure monitoring-based analysis of long-term outcomes for kidney disease progression. Sci Rep. 2019 Dec 17;9(1):19296. doi: 10.1038/s41598-019-55732-4. PMID 31848394
- [Background] Kanno A, Kikuya M, Asayama K, Satoh M, Inoue R, Hosaka M, Metoki H, Obara T, Hoshi H, Totsune K, Sato T, Taguma Y, Sato H, Imai Y, Ohkubo T. Night-time blood pressure is associated with the development of chronic kidney disease in a general population: the Ohasama Study. J Hypertens. 2013 Dec;31(12):2410-7. doi: 10.1097/HJH.0b013e328364dd0f. PMID 24029869
- [Background] Minutolo R, Agarwal R, Borrelli S, Chiodini P, Bellizzi V, Nappi F, Cianciaruso B, Zamboli P, Conte G, Gabbai FB, De Nicola L. Prognostic role of ambulatory blood pressure measurement in patients with nondialysis chronic kidney disease. Arch Intern Med. 2011 Jun 27;171(12):1090-8. doi: 10.1001/archinternmed.2011.230. PMID 21709109
- [Background] Mojon A, Ayala DE, Pineiro L, Otero A, Crespo JJ, Moya A, Boveda J, de Lis JP, Fernandez JR, Hermida RC; Hygia Project Investigators. Comparison of ambulatory blood pressure parameters of hypertensive patients with and without chronic kidney disease. Chronobiol Int. 2013 Mar;30(1-2):145-58. doi: 10.3109/07420528.2012.703083. Epub 2012 Oct 25. PMID 23181690
- [Background] Rahman M, Wang X, Bundy JD, Charleston J, Cohen D, Cohen J, Drawz PE, Ghazi L, Horowitz E, Lash JP, Schrauben S, Weir MR, Xie D, Townsend RR; CRIC Study Investigators. Prognostic Significance of Ambulatory BP Monitoring in CKD: A Report from the Chronic Renal Insufficiency Cohort (CRIC) Study. J Am Soc Nephrol. 2020 Nov;31(11):2609-2621. doi: 10.1681/ASN.2020030236. Epub 2020 Sep 24. PMID 32973085
- [Background] Stergiou GS, Palatini P, Parati G, O'Brien E, Januszewicz A, Lurbe E, Persu A, Mancia G, Kreutz R; European Society of Hypertension Council and the European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement. J Hypertens. 2021 Jul 1;39(7):1293-1302. doi: 10.1097/HJH.0000000000002843. No abstract available. PMID 33710173
- [Background] Wang C, Zhang J, Liu X, Li C, Ye Z, Peng H, Chen Z, Lou T. Reversed dipper blood-pressure pattern is closely related to severe renal and cardiovascular damage in patients with chronic kidney disease. PLoS One. 2013;8(2):e55419. doi: 10.1371/journal.pone.0055419. Epub 2013 Feb 5. PMID 23393577